CLINICAL TRIAL: NCT00731536
Title: A Retrospective Review of Reports of Hepatosplenic T-cell Lymphoma in the Dutch National Database of Pathology (Pathologisch-Anatomisch Landelijk Geautomatiseerd Archief [PALGA]), a Database of Pathology Results for The Netherlands
Brief Title: Observational Study on the Occurrence of Hepatosplenic T-cell Lymphoma in Patients of Netherlands
Status: Completed | Type: Observational
Sponsor: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015394; C0168Z06 (Other: Centocor, Inc.)
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Hepatosplenic T-cell Lymphoma
Keywords: Hepatosplenic T-cell Lymphoma; Remicade; Infliximab; Dutch national database of pathology; PALGA; Autoimmune disease; Non-Hodgkin lymphoma
MeSH Terms: conditions — Autoimmune Diseases; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Hepatosplenic T-cell Lymphoma (HSTCL)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. Medical records of patients with the diagnosis of HSTCL in the PALGA database will be analyzed.

SUMMARY:
The purpose of this study is to examine reports of the cancer called hepatosplenic T-cell lymphoma (HSTCL) in the Dutch National Database of Pathology (Pathologisch-Anatomisch Landelijk Geautomatiseerd Archief or PALGA) during the years 1995 to 2008.

DETAILED DESCRIPTION:
This is a observational, retrospective (a study in which the participants are identified and then followed backward in time, for the outcome of the study) study. In this study review of all reports of possible cases of hepatosplenic T-cell lymphoma (HSTCL) that were identified within the PALGA database of pathology results for The Netherlands from 1995 to 2008. All patients whose information is contained within the PALGA database were prescribed treatments by a physician on the basis of usual clinical practice or may have received other treatments, including experimental drugs, while participating in an interventional clinical study. The identified data on each of the patients with reports of HSTCL will be collected from the pathologist(s) who prepared the report and from the physician(s) who treated the patient at the time of diagnosis.

ELIGIBILITY:
Inclusion Criteria:

- Patients diagnosed with HSTCL in the Dutch National Database of Pathology (Pathologisch-Anatomisch Landelijk Geautomatiseerd Archief) database during the years 1995 to 2008

Exclusion Criteria:

- Patients who are not diagnosed with HSTCL

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hepatosplenic T-cell Lymphoma (HSTCL).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with diagnosis of Hepatosplenic T-cell Lymphoma (HSTCL) | 1 year
  Evaluation of the occurrence of the diagnosis of HSTCL among patients with pathology reports in the Pathologisch-Anatomisch Landelijk Geautomatiseerd Archief (PALGA) database during the years 1995 to 2008.

SECONDARY OUTCOMES:
Number of patients with HSTCL that are present in the population of The Netherlands | 1 year
  Number of cases with HSTCL will be used to evaluate the prevalence.
Number of newly diagnosed patients with HSTCL that are present in the population of The Netherlands | 1 year
  Number of newly diagnosed patients with HSTCL will be used to evaluate the incidence of HSTCL.
Number of newly diagnosed patients with HSTCL that are present in the population of The Netherlands prior to and after the availability of infliximab | 1 year
  Number of newly diagnosed patients with HSTCL will be used to evaluate the incidence of HSTCL prior to and after the availability of infliximab.
Data collection for factors associated with the diagnosis of HSTCL | 1 year
  Data collection will include HSCTL diagnosis, diseases and medical/surgical conditions, cytogenetic data, and demographic data.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Ortho Biotech Services, L.L.C. Clinical Trial, Study Director — Centocor Ortho Biotech Services, L.L.C.
Locations (10):
- Netherlands (10):
  - Alkmaar
  - Amsterdam
  - Amsterdam-Zuidoost
  - Eindhoven
  - Groningen
  - Nijmegen
  - Oss
  - Rotterdam
  - Utrecht
  - Winschoten